CLINICAL TRIAL: NCT00739076
Title: Pain Control After Trauma
Acronym: VRHTrauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, David Patterson, PhD. ABPP. Professor, National Institute of General Medical Sciences (NIGMS)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30359-G; R01GM042725-09A1 (NIH)
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Virtual Reality Hypnosis
  Interventions: Behavioral: Virtual Reality
- 2 (Experimental): Virtual Reality Distraction
  Interventions: Behavioral: Virtual Reality
- 3 (Experimental): Standard treatment.
  Interventions: Behavioral: Virtual Reality

INTERVENTIONS:
Behavioral: Virtual Reality — Using Virtual Reality for pain control

SUMMARY:
Using Virtual Reality as a form of pain control for trauma patients.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effectiveness of virtual reality (a form of distraction) in order to reduce patients' pain from trauma.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 12 years
* Compliant and able to complete questionnaires
* Hospitalization for internal injuries requiring a laparotomy or for orthopedic injuries (closed long bone or calcaneus fractures).
* A minimum of 3 days hospitalization
* No history of psychiatric (DSM-IV-R Axis I) disorder
* Not demonstrating delirium, psychosis or any form of Organic Brain Disorder
* Able to communicate verbally
* Able to take oral medications
* Baseline pain level of >=5/10
* English-speaking

Exclusion Criteria:

* Age less than 12 years
* Not capable of indicating pain intensity
* Not capable of filling out study measures
* Hospitalization of less than 3 days
* Evidence of traumatic brain injury
* History of psychiatric (DSM-IV-R Axis I) disorder as evidenced in the admitting RN and MD admission notes.
* Demonstrating delirium, psychosis or any form of Organic Brain Disorder and associated memory problems.
* Unable to communicate orally.
* Unable to take oral medications
* History of sig. cardiac, endocrine, neurologic, metabolic, respiratory, gastrointestinal or genitourinary impairment
* Receiving prophylaxis for alcohol or drug withdrawal
* Developmental disability
* Mini-mental status score of greater than 20 in patients older than 80 years or suspected of cognitive deficits
* Non-English Speaking
* Extreme susceptibility to motion sickness
* Seizure history

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2007-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain and Anxiety | up to 3 times a day

CONTACTS AND LOCATIONS:
Overall Officials: David R Patterson, Ph.D, Principal Investigator — University of Washington
Locations (1):
- University of Washington; Harborview Medical Center, Seattle, Washington, United States